CLINICAL TRIAL: NCT04948281
Title: The Effects of Joint Infection Following Arthroscopic Single-bundle ACL Reconstruction With Autologous Hamstring: a Retrospective Matched Cohort Study
Brief Title: Joint Infection Following ACL Reconstruction
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017332
Record Dates: First submitted 2021-06-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection Group: A group of joint infection patients after arthroscopic ACL reconstruction surgery , diagnose was made according to American CDC criteria of joint infection
  Interventions: Other: no intervention
- Control Group: A group of patients which were matched to infections group retrospectively one-to-three who did not sustain any kind of infection after ACL reconstruction.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study was conducted to analyze the effect of joint infection on the bone tunnel, graft and articular cartilage following arthroscopic single-bundle anterior cruciate ligament (ACL) reconstruction with autologous hamstring, to summarize the features of MR findings after joint infection, and to correlate these findings with their possible factors.

DETAILED DESCRIPTION:
A retrospective matched cohort study was performed in 26 patients who underwent arthroscopic single-bundle ACL reconstruction with hamstring graft and developed postoperative joint infection in our institute from January 2002 to December 2017. They were matched 1:3 to patients who did not sustain joint infection after ACL reconstruction. MR scan was collected at the time of follow-up. Bone tunnel enlargement at tunnel aperture, midsection and exit of tibial and femoral tunnel was carefully assessed. Graft signal-to-noise quotient (SNQ) on MRI was calculated to evaluate graft maturity. Cartilage morphology was graded using Whole Organ Magnetic Resonance Imaging Score. A generalized linear mixed model was applied to analyze the effect of joint infection on the bone tunnel, graft and articular cartilage.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 to 50 years;
* Underwent single-bundle ACL reconstruction with autologous hamstring;
* Had valid follow-up magnetic resonance imaging (MRI) at least 1 year after surgery

Exclusion Criteria:

* Concomitant ligament injury which need surgical repair;
* Delayed onset of postoperative joint infection (>3 months after surgery).

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population were from 20549 arthroscopic ACL reconstruction surgeries in our institute between January 2002 to December 2017.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Tunnel enlargement | 1 year after operation/infection
  A 3.0T MRI unit (General Electric Healthcare) with an 8-channel coil was used for measurement. Anteroposterior and lateromedial diameter at tunnel aperture, midsection and exit of tibial and femoral tunnel (demonstrated as TTa, TTm, TTe, FTa, FTm, FTe) was measured on T1-weighted images (in millimeters)
Graft signal intensity | 1 year after operation/infection
  Proton Density weighted fat suppressed turbo-spin echo (PD-TSE-FS) sequence was taken to calculate the SNQof the graft. Graft signal intensity was measured at proximal, middle and distal end of the graft.
Cartilage morphology | 1 year after operation/infection
  The cartilage morphology at surgery was assessed using Outerbridge classification for chondral lesion and recorded in operation note. cartilage morphology was assessed according to the Whole-organ magnetic scoring system (WORMS) of the knee on sagittal and axial T2-weighted FSE images.

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided